CLINICAL TRIAL: NCT05538286
Title: Transcranial Ultrasound Via Sonolucent Cranioplasty After Minimally Invasive Intracerebral Hemorrhage Evacuation
Acronym: TUSC MIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Christopher P Kellner, Associate Professor, Department of Neurosurgery, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-21-01878
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Transcranial Ultrasound With Sonolucent Cranioplasty; TUSC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- transcranial ultrasonography through sonolucent cranioplasty (Experimental): All surgical procedures and implants in this protocol are standard of care.
  Interventions: Device: ClearFit implant; Procedure: transcranial ultrasonography through sonolucent cranioplasty

INTERVENTIONS:
Device: ClearFit implant — The ClearFit implant is an FDA cleared implant in regular use in the United States. The ClearFit implant and other PMMA cranioplasty implants manufactured by Longeviti have been reported to be safe and effective as cranial implants that permit transcranial ultrasound to be performed. The PMMA cranioplasty implant (Longeviti Neuro Solutions, Hunt Valley, MD) is clear, sonolucent, and was recently shown to be safe and effective in transcranial ultrasonography for bypass patency assessment. The ClearFit cranioplasty being used in this study is industry standard of care.
Procedure: transcranial ultrasonography through sonolucent cranioplasty — The implantation of the ClearFit PMMA sonolucent implant permits TUSC to be performed at the bedside for patients in both the in-patient and outpatient settings. While the patient is an inpatient, the clinical or research teams will attempt to perform TUSC within 1 hour of neuroimaging if that neuroimaging is performed at a time when a trained ultrasound operator is present.
  Other Names: TUSC

SUMMARY:
Postoperative rebleeding is a major limitation of surgical evacuation for intracerebral hemorrhage (ICH). While computed tomography (CT) is the standard of care for postoperative hematoma cavity monitoring, CT requires significant physical and financial costs. Studies have demonstrated varying degrees of efficacy when using transcranial ultrasound to measure ICH volume. Recently, synthetic implants for cranioplasty have been shown to be safe and sonolucent. This study aims to evaluate the ability of transcranial ultrasound with sonolucent cranioplasty (TUSC) to detect and quantify bleeding in postoperative ICH patients.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) accounts for over 2 million strokes annually. ICH is the most devastating subtype of stroke, with a 1-year mortality rate of up to 50% and a 6-month survivor disability rate of up to 88%. Large-scale multicenter trials including STICH, STICH II, and MISTIE III demonstrated that surgical evacuation did not appear to improve long term functional outcome. Smaller studies and sub-group analyses have suggested that some forms of minimally invasive ICH evacuation may benefit specific patients. Postoperative rebleeding after surgical evacuation of ICH occurs in 5-40% and remains a major limitation to the efficacy and widespread adoption of this treatment strategy. Therefore, rapid assessment, detection, and management of postoperative bleeding is critical to maximize functional recovery after surgical evacuation.

The standard of care for postoperative hematoma cavity monitoring is computed tomography (CT). However, repeat CTs to assess patients with ICH incur health and financial cost including time and personnel to bring the patient to scan, risk of dislodging lines or drains, radiation dosing, and financial cost as well as others. Studies have demonstrated varying degrees of efficacy when using transcranial ultrasound to measure ICH volume. Recently, synthetic implants for cranioplasty have been shown to be safe and sonolucent. This study aims to evaluate the ability of transcranial ultrasound with sonolucent cranioplasty (TUSC) to detect and quantify bleeding in postoperative ICH patients.

In this prospective study, postoperative ICH patients will undergo cranioplasty with a sonolucent polymethyl methacrylate implant and serial monitoring via TUSC. Whenever a CT is performed during business hours, TUSC will be performed within 2 hours by a neurointensivist trained in point-of-care transcranial ultrasound (TCUS). Imaging will be reviewed by two independent neuroimaging experts. Additional secondary outcomes will include occurrence of serious adverse events, detection of intraventricular hemorrhage, and cost of care when compared to CT.

This work has the potential to significantly improve clinical management of ICH. This study will provide the safety and feasibility data necessary to guide future clinical research. ICH detection and volumetry are critical to patient care and prognostication. This point-of-care testing enables neurosurgeons to serially monitor patients to ensure that they receive timely, appropriate care.

ELIGIBILITY:
Inclusion criteria:

* Presence of spontaneous supratentorial ICH ≥20 mL
* Age ≥18 years
* National Institute of Health Stroke Scale (NIHSS) score ≥6
* GCS score 5-15 at presentation
* Undergoing minimally invasive intracerebral hemorrhage evacuation with sonolucent cranioplasty or hemicraniectomy with sonolucent cranioplasty

Exclusion criteria:

* Secondary cause for the ICH, such as an underlying vascular malformation (cavernous malformation, arteriovenous malformation, etc.), aneurysm, neoplasm, hemorrhagic transformation of an underlying ischemic infarct; or venous infarct
* History of osteomyelitis
* History of skull neoplasm
* History of comminuted skull fractures
* Infratentorial hemorrhage
* Midbrain extension/involvement
* Coagulopathy defined as INR > 1.4, elevated aPTT, or concurrent use of direct oral anticoagulants or low molecular weight heparin at ICH onset; known hereditary or acquired hemorrhagic diathesis; coagulation factor deficiency; platelet count < 100x103cells/mm3, or known platelet dysfunction
* Inability to obtain consent from patient or appropriate surrogate (for patients without capacity)
* Evidence of active infection indicated by fever ≥ 100.7F and/or open draining wound at the time of enrolment
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 1 year
* Based on investigator's judgment, the patient does not have the necessary mental capacity to participate or is unwilling to comply with the protocol follow-up appointment schedule
* Active drug or alcohol abuse that, in the opinion of the site investigator, would interfere with adherence to study enrolments
* Pre-existing DNR/DNI status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The presence of intracerebral hemorrhage | at 6 months
  Accuracy of TUSC via ClearFit to detect the presence or absence of postoperative intracerebral hemorrhage compared to CT.

SECONDARY OUTCOMES:
Serious Adverse Events related to ClearFit or TUSC | at 6 months
  Serious Adverse Events related to ClearFit or TUSC
Accuracy of TUSC to detect intraventricular hemorrhage | at 6 months
  Accuracy of TUSC to detect intraventricular hemorrhage compared to CT. Detection of intraventricular hemorrhage will be a categorical variable [present, absent].
TUSC/CT ratio for distance between lateral ventricle frontal horns | at 6 months
  TUSC/CT ratio to measure distance between lateral ventricle frontal horns.
TUSC/CT ratio for midline shift | at 6 months
  TUSC/CT ratio to measure midline shift
Accuracy of TUSC to detect hydrocephalus | at 6 months
  Detection of hydrocephalus will be a categorical variable based on ventricle morphology and size [present, absent]
Cost of TUSC | at 6 months
  Cost of TUSC versus standard of care imaging (CT or MRI)
Reimbursement rates for TUSC | at 6 months
  Reimbursement rates for TUSC as a point of care examination in the ICU and outpatient clinic

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Kellner, MD, Principal Investigator — Mount Sinai Health System Department of Neurosurgery
Locations (1):
- Mount Sinai Health System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
In order to minimize any privacy risks to the patients participating, IPD data will not be shared.

REFERENCES:
- [Background] Niesen WD, Schlaeger A, Bardutzky J, Fuhrer H. Correct Outcome Prognostication via Sonographic Volumetry in Supratentorial Intracerebral Hemorrhage. Front Neurol. 2019 May 8;10:492. doi: 10.3389/fneur.2019.00492. eCollection 2019. PMID 31133979
- [Background] Krishnamurthi RV, Feigin VL, Forouzanfar MH, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson LM, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, Risk Factors Study 2010 (GBD 2010); GBD Stroke Experts Group. Global and regional burden of first-ever ischaemic and haemorrhagic stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet Glob Health. 2013 Nov;1(5):e259-81. doi: 10.1016/S2214-109X(13)70089-5. Epub 2013 Oct 24. PMID 25104492
- [Background] Kellner CP, Song R, Pan J, Nistal DA, Scaggiante J, Chartrain AG, Rumsey J, Hom D, Dangayach N, Swarup R, Tuhrim S, Ghatan S, Bederson JB, Mocco J. Long-term functional outcome following minimally invasive endoscopic intracerebral hemorrhage evacuation. J Neurointerv Surg. 2020 May;12(5):489-494. doi: 10.1136/neurintsurg-2019-015528. Epub 2020 Jan 8. PMID 31915207
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Background] Morgenstern LB, Demchuk AM, Kim DH, Frankowski RF, Grotta JC. Rebleeding leads to poor outcome in ultra-early craniotomy for intracerebral hemorrhage. Neurology. 2001 May 22;56(10):1294-9. doi: 10.1212/wnl.56.10.1294. PMID 11376176
- [Background] Delcourt C, Huang Y, Arima H, Chalmers J, Davis SM, Heeley EL, Wang J, Parsons MW, Liu G, Anderson CS; INTERACT1 Investigators. Hematoma growth and outcomes in intracerebral hemorrhage: the INTERACT1 study. Neurology. 2012 Jul 24;79(4):314-9. doi: 10.1212/WNL.0b013e318260cbba. Epub 2012 Jun 27. PMID 22744655
- [Background] Flores AR, Srinivasan VM, Seeley J, Huggins C, Kan P, Burkhardt JK. Safety, Feasibility, and Patient-Rated Outcome of Sonolucent Cranioplasty in Extracranial-Intracranial Bypass Surgery to Allow for Transcranioplasty Ultrasound Assessment. World Neurosurg. 2020 Dec;144:e277-e284. doi: 10.1016/j.wneu.2020.08.114. Epub 2020 Aug 20. PMID 32827747
- [Background] Kellner CP, Song R, Ali M, Nistal DA, Samarage M, Dangayach NS, Liang J, McNeill I, Zhang X, Bederson JB, Mocco J. Time to Evacuation and Functional Outcome After Minimally Invasive Endoscopic Intracerebral Hemorrhage Evacuation. Stroke. 2021 Aug;52(9):e536-e539. doi: 10.1161/STROKEAHA.121.034392. Epub 2021 Jun 24. PMID 34424739
- [Background] Fernando SM, Qureshi D, Talarico R, Dowlatshahi D, Sood MM, Smith EE, Hill MD, McCredie VA, Scales DC, English SW, Rochwerg B, Tanuseputro P, Kyeremanteng K. Short- and Long-term Health Care Resource Utilization and Costs Following Intracerebral Hemorrhage. Neurology. 2021 Aug 10;97(6):e608-e618. doi: 10.1212/WNL.0000000000012355. Epub 2021 Jun 9. PMID 34108269
- [Background] Hadley C, North R, Srinivasan V, Kan P, Burkhardt JK. Elective Sonolucent Cranioplasty for Real-Time Ultrasound Monitoring of Flow and Patency of an Extra- to Intracranial Bypass. J Craniofac Surg. 2020 May/Jun;31(3):622-624. doi: 10.1097/SCS.0000000000006225. PMID 32149973